CLINICAL TRIAL: NCT02764125
Title: Efficacy and Safety of ODM-104 Compared to a Standard Combination (Stalevo®); a Randomized Double-blind, Crossover Proof-of-concept Study in Patients With Parkinson's Disease and End-of-dose Wearing-off
Brief Title: Efficacy and Safety Proof of Concept Study in Patients With Parkinson's Disease and End-of-dose Wearing-off (COMPOC)
Acronym: COMPOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3112004
Record Dates: First submitted 2016-01-13; First posted 2016-05-06 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Wearing-off
MeSH Terms: conditions — Parkinson Disease | interventions — Stalevo; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stalevo (Active Comparator): levodopa/carbidopa/entacapone
  Interventions: Drug: Stalevo
- levodopa MR (Experimental): Levodopa MR/carbidopa/ODM-104
  Interventions: Drug: levodopa MR

INTERVENTIONS:
Drug: Stalevo — levodopa/carbidopa/entacapone
  Other Names: levodopa/carbidopa/entacapone
  Arms: Stalevo
Drug: levodopa MR — levodopa MR/carbidopa/ODM-104
  Other Names: levodopa MR/carbidopa/ODM-104
  Arms: levodopa MR

SUMMARY:
This will be a randomised, crossover, double-blind, double-dummy, active-controlled, multicentre, phase II proof-of-concept study in Parkinson's Disease (PD) patients with end-of-dose wearing-off (motor fluctuations).

DETAILED DESCRIPTION:
This will be a randomised, crossover, double-blind, double-dummy, active-controlled, multicentre, phase II proof-of-concept study in PD patients with end-of-dose wearing-off (motor fluctuations).

In a 2-period crossover design the subjects will receive ODM-104/levodopa/ carbidopa or Stalevo during the different study periods in a randomised order. There will be a screening period, 2 treatment periods and a post-treatment period, altogether 7 scheduled visits: a screening visit, a baseline visit, 4 visits during the treatment periods (i.e. 2 visits/each period), and an end-of-study visit. Unscheduled visits may be performed during the first 2 weeks of each treatment period, if there is a need to adjust the levodopa strength. The total study duration will be 10-15 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (IC) obtained.
* Male or female patients with idiopathic PD according to the UK brain bank criteria with end-of-dose wearing-off (motor fluctuations).
* Hoehn and Yahr stage 2-4 performed during the ON-state.
* At least 2 hours of OFF-time on each day (measured by the ON/OFF diary) on 3 consecutive days at the end of the screening period just before the baseline visit (visit 1).
* Treatment with 4-8 daily doses of levodopa/AADC inhibitor, either combined with entacapone (levodopa/AADC inhibitor combined with Comtess/Comtan or as Stalevo) or without entacapone, with a total daily levodopa dose from > 400 mg to ≤ 1200 mg with entacapone, or from > 400 mg to ≤ 1400 mg without entacapone. One evening dose of controlled release formulation, 1 morning dose of soluble levodopa/AADC inhibitor, or both, as needed are allowed.
* Unchanged levodopa/AADC inhibitor with or without entacapone, and other antiparkinsonian medication (dopamine agonists, monoamine oxidase [MAO] B inhibitor, amantadine and/or anticholinergics with doses recommended by the manufacturer), if any, for at least 4 weeks before the screening visit.
* Age of 30 years or above.

Exclusion Criteria:

* Secondary or atypical Parkinsonism.
* Current use of tolcapone or opicapone (within 4 weeks before the screening visit).
* Previous tolerability problems with entacapone, tolcapone or opicapone.
* Concomitant treatment with apomorphine, MAO-A inhibitors or non-selective MAO inhibitors (within 4 weeks before the screening visit).
* Concomitant treatment with drugs having antidopaminergic action including alpha-methyldopa, reserpine and antipsychotic drugs (also D2 receptor blocking antiemetics except domperidone). As an exception to prohibit use of antipsychotic drugs, 1 evening dose of an atypical antipsychotic is allowed.
* Use of concomitant medicine which is predominantly metabolised by CYP3A4 and which has a narrow therapeutic window such as ergot alkaloids, carbamazepine, cyclosporin, macrolides (sirolimus and tacrolimus), quinidine or fentanyl.
* Current use of warfarin (within 4 weeks before the screening visit).
* Inability to refrain from use of any iron preparations during the study.
* Disabling dyskinesias.
* Problematic hallucinations within 3 months before the screening visit.
* Symptomatic orthostatic hypotension.
* Current dementia (Mini Mental State Examination [MMSE] score < 26).
* Problematic impulse control disorders (ICDs), such as pathological gambling, hypersexuality or compulsive shopping within 6 months before the screening visit.
* History of neuroleptic malignant syndrome (NMS), non-traumatic rhabdomyolysis, or both.
* Any neurosurgical intervention for the treatment of PD, including deep brain stimulation (DBS).
* Narrow-angle glaucoma or pheochromocytoma.
* Any active malignant cancer.
* Clinically significant cardiovascular (e.g. ischaemic heart disease, ventricular or supraventricular arrhythmias), pulmonary, GI (e.g. inflammatory bowel disease), hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part into the study.
* Alanine aminotransferase or aspartate aminotransferase > 1.25 x upper limit of normal (ULN) at screening.
* Any other abnormal value of laboratory, vital signs or ECG (such as QTcF prolongation ≥ 450 ms) that may in the opinion of the investigator interfere with the interpretation of the study results or cause health risk for the subject if he/she takes part into the study.
* Female patients of childbearing potential (i.e. menstruating or less than 2 years postmenopausal).
* Patients with pre-planned surgery requiring hospitalisation during the study.
* Known hypersensitivity to active substances or to any of the excipients of the study treatments.
* Blood donation or loss of significant amount of blood within 60 days before screening visit.
* Participation in a drug study within 60 days before the first treatment period.
* Any other condition that in the opinion of the investigator would interfere with the interpretation of the study results or constitute a health risk for the subject if he/she takes part into the study.
* Failure to demonstrate acceptable/appropriate use of the ON/OFF diary despite adequate training during the screening visit.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Duration of daily OFF-time (measured by Hauser ON/OFF-diary) | 3 consecutive days in the end of both periods compared to 3 consecutive days prior the baseline visit.
  OFF-time (time when the patient does not experience a positive response to medication between the study drug intake) measured from the Hauser ON/OFF-diary that patient has filled in (24 hour clock) for 3 days prior to baseline visit and at the end of both treatment periods.

SECONDARY OUTCOMES:
Switching patients from their regular levodopa treatment to planned new treatment. | two 4 weeks study periods
  To explore how to switch patients on levodopa/aromatic amino acid decarboxylase (AADC) inhibitor or levodopa/AADC inhibitor + entacapone directly to ODM-104 in combination with MR levodopa and carbidopa by evaluating how much adjustments to levodopa strengths need to be done and if there is difference between the two treatment groups.
Determination of sample size | two 4 weeks study periods
  To determine the effect size for phase III planning if the difference between the two study treatment groups with this amount of patients can be shown.
To show adequate Parkinson's Disease symptom control with the new treatment | two 4 weeks study periods
  To study levodopa daily dose and dosing frequency of the combination to see if Parkinson's disease symptoms are adequately controlled with study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aila Holopainen, MSc, Study Director — Orion Corporation, Orion Pharma, Development
Locations (4):
- Clinical Research Services Turku CRST, Turku, Finland
- Study Coordinating Investigator, Harleshausen, Kassel, Germany
- Semmelweis Egyetem Neurológiai Klinika, Budapest, Hungary
- Investigator, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No